CLINICAL TRIAL: NCT02670941
Title: Aromatherapy for Management of Chemotherapy-induced Symptoms
Brief Title: Aromatherapy for Chemotherapy-induced Symptoms
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Slow accrual; Received grant funding for a similar but different study.
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Julie Ryan, Assistant Professor of Dermatology, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSRB57258
Record Dates: First submitted 2016-01-15; First posted 2016-02-02 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Chemotherapy Symptoms
Keywords: aromatherapy; chemotherapy; ginger; lavender; orange; jojoba; essential oils; cancer
MeSH Terms: conditions — Neoplasms | interventions — ginger extract; lavender oil; jojoba wax

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Ginger (Experimental): Subjects will use the aromatherapy inhalers through three chemotherapy treatment cycles (i.e., Study Cycle 1, Study Cycle 2, and Study Cycle 3). During each Study Cycle, subjects will start the aromatherapy inhaler on the day before the start of their chemotherapy treatment cycle (Day 0) and continue using the inhaler for the next six consecutive days (Day 1-Day 6), including the day he/she starts their chemotherapy treatment cycle. The subjects will remove the cover of the aromatherapy inhaler, place the aromatherapy inhaler under their nose and inhale three times with deep breathing (i.e., three sniffs). After use, the inhaler should be capped to minimize dispersal of the scent. Subjects will take 3 sniffs of the aromatherapy inhaler four times daily (morning, noon, evening, bedtime).
  Interventions: Drug: Ginger
- Lavender (Experimental): Subjects will use the aromatherapy inhalers through three chemotherapy treatment cycles (i.e., Study Cycle 1, Study Cycle 2, and Study Cycle 3). During each Study Cycle, subjects will start the aromatherapy inhaler on the day before the start of their chemotherapy treatment cycle (Day 0) and continue using the inhaler for the next six consecutive days (Day 1-Day 6), including the day he/she starts their chemotherapy treatment cycle. The subjects will remove the cover of the aromatherapy inhaler, place the aromatherapy inhaler under their nose and inhale three times with deep breathing (i.e., three sniffs). After use, the inhaler should be capped to minimize dispersal of the scent. Subjects will take 3 sniffs of the aromatherapy inhaler four times daily (morning, noon, evening, bedtime).
  Interventions: Drug: Lavender
- Orange (Experimental): Subjects will use the aromatherapy inhalers through three chemotherapy treatment cycles (i.e., Study Cycle 1, Study Cycle 2, and Study Cycle 3). During each Study Cycle, subjects will start the aromatherapy inhaler on the day before the start of their chemotherapy treatment cycle (Day 0) and continue using the inhaler for the next six consecutive days (Day 1-Day 6), including the day he/she starts their chemotherapy treatment cycle. The subjects will remove the cover of the aromatherapy inhaler, place the aromatherapy inhaler under their nose and inhale three times with deep breathing (i.e., three sniffs). After use, the inhaler should be capped to minimize dispersal of the scent. Subjects will take 3 sniffs of the aromatherapy inhaler four times daily (morning, noon, evening, bedtime).
  Interventions: Drug: Orange
- Jojoba (Placebo Comparator): Subjects will use the aromatherapy inhalers through three chemotherapy treatment cycles (i.e., Study Cycle 1, Study Cycle 2, and Study Cycle 3). During each Study Cycle, subjects will start the aromatherapy inhaler on the day before the start of their chemotherapy treatment cycle (Day 0) and continue using the inhaler for the next six consecutive days (Day 1-Day 6), including the day he/she starts their chemotherapy treatment cycle. The subjects will remove the cover of the aromatherapy inhaler, place the aromatherapy inhaler under their nose and inhale three times with deep breathing (i.e., three sniffs). After use, the inhaler should be capped to minimize dispersal of the scent. Subjects will take 3 sniffs of the aromatherapy inhaler four times daily (morning, noon, evening, bedtime).
  Interventions: Drug: Jojoba

INTERVENTIONS:
Drug: Ginger — The ginger oil (GIN-106) was steam distilled from fresh ginger grown in Madagascar. The ginger oil contains 64.23% sesquiterpenes, 18.5% monoterpenes, and 3.28% aldehydes. The aroma of ginger is described as spicy, sweet, and warm.
  Arms: Ginger
Drug: Lavender — The lavender oil (LAV-110) was steam distilled from lavender grown in Kashmir Valley in India. The lavender oil contains 53.22% esters, 31.86% monoterpenols, and 4.88% oxides. The aroma of lavender is described as floral, fresh, herbaceous, and sweet.
  Arms: Lavender
Drug: Orange — The orange oil (ORG-114) was cold-pressed and steam distilled from oranges in South Africa. The orange oil contains 97.21% monoterpenes, 0.73% aldehydes, and 0.7% monoterpenols. The aroma of orange is described as citrus, fresh, fruity, and sweet.
  Arms: Orange
Drug: Jojoba — The jojoba oil is certified organic and pesticide-free pure oil. Jojoba has a mild scent and can be used as a "fixative" for other essential oils.
  Arms: Jojoba

SUMMARY:
The rationale behind the proposed study is to determine the initial effectiveness of aromatherapy in relief of commonly reported symptoms in cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
The proposed study is an exploratory trial to evaluate the use of aromatherapy for symptom management in patients undergoing chemotherapy. The investigators will accrue 120 adult cancer subjects undergoing chemotherapy in a initial efficacy study to determine the effectiveness of three different aromatherapies (ginger, lavender, or orange) on chemotherapy-related symptoms (nausea, vomiting, pain, anxiety, sleep difficulties, fatigue, and lack of appetite) compared to placebo (i.e., jojoba). All subjects will be randomized to one of the four arms for symptom management during three different chemotherapy cycles. The investigators will examine the incidence and severity of the seven symptoms at each chemotherapy cycle. The preliminary data from this study will elucidate the relationships between certain aromatherapies and specific symptom relief, which can be further evaluated in a larger confirmatory study of subjects undergoing chemotherapy or other types of cancer treatment. This study will provide clinical evidence regarding the incorporation of aromatherapy into cancer patient care.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adults between the ages of 21 to 89 years of age with diagnosis of cancer and be scheduled to receive at least three more cycles of chemotherapy.
* Subjects must have had at least one chemotherapy cycle in their current prescribed course and have at least three additional chemotherapy cycles planned.
* Day 1 of each chemotherapy cycle must be separated from Day 1 of the next chemotherapy cycles by at least 12 days.
* All chemotherapy regimens are eligible.
* Any number of chemotherapy administrations per week during a chemotherapy treatment cycle is allowed.
* Subjects agree to discontinue any current aromatherapy usage and only use the study aromatherapy for symptom management during the course of the study. NOTE: Patients can continue to use scented soaps, lotions, shampoos, body sprays, perfume/cologne, candles, or air fresheners that they regularly use.
* Subjects must be able to read and understand English, as well as provide informed consent in order to participate in this study.

Exclusion Criteria:

* Subjects < 21 years old or > 89 years old are not eligible for participation in this study at the University of Rochester.
* Pregnant females are ineligible for the study because pregnancy is a contraindication for chemotherapy and exposure to essentials oils.
* Subjects who are chemotherapy-naïve are ineligible.
* Subjects with more than four weeks between chemotherapy treatment cycles are not eligible.
* Concurrent radiation therapy or interferon treatment is not allowed.
* Subjects that have used or are currently using aromatherapy inhalation for symptom management are not eligible.
* Subjects with any known allergy to ginger, lavender, orange, citrus of any kind, jojoba, or essential oils.

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-01; Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

PRIMARY OUTCOMES:
Mean change in severity in symptoms | up to 11 weeks
  Subjects will complete a self-report Symptom Inventory Diary during each Study Cycle starting at Day 0 and continuing to Day 6. Subjects will rate the severity of seven symptoms (nausea, vomiting, pain, anxiety/distress, sleep difficulties, fatigue, and lack of appetite) using a 0-10 numeric rating scale, with 10 indicating a higher severity, in daily diary format.

SECONDARY OUTCOMES:
change in mean peak severity for nausea across all three cycles | up to 11 weeks
  Subjects will complete a self-report Symptom Inventory Diary during each Study Cycle starting at Day 0 and continuing to Day 6. Subjects will rate the severity of seven symptoms (nausea, vomiting, pain, anxiety/distress, sleep difficulties, fatigue, and lack of appetite) using a 0-10 numeric rating scale, with 10 indicating a higher severity, in daily diary format.
change in mean peak severity for vomiting across all three cycles | up to 11 weeks
  Subjects will complete a self-report Symptom Inventory Diary during each Study Cycle starting at Day 0 and continuing to Day 6. Subjects will rate the severity of seven symptoms (nausea, vomiting, pain, anxiety/distress, sleep difficulties, fatigue, and lack of appetite) using a 0-10 numeric rating scale, with 10 indicating a higher severity, in daily diary format.
change in mean peak severity for anxiety/distress across all three cycles | up to 11 weeks
  Subjects will complete a self-report Symptom Inventory Diary during each Study Cycle starting at Day 0 and continuing to Day 6. Subjects will rate the severity of seven symptoms (nausea, vomiting, pain, anxiety/distress, sleep difficulties, fatigue, and lack of appetite) using a 0-10 numeric rating scale, with 10 indicating a higher severity, in daily diary format.
change in mean peak severity for pain across all three cycles | up to 11 weeks
  Subjects will complete a self-report Symptom Inventory Diary during each Study Cycle starting at Day 0 and continuing to Day 6. Subjects will rate the severity of seven symptoms (nausea, vomiting, pain, anxiety/distress, sleep difficulties, fatigue, and lack of appetite) using a 0-10 numeric rating scale, with 10 indicating a higher severity, in daily diary format.
change in mean peak severity for fatigue across all three cycles | up to 11 weeks
  Subjects will complete a self-report Symptom Inventory Diary during each Study Cycle starting at Day 0 and continuing to Day 6. Subjects will rate the severity of seven symptoms (nausea, vomiting, pain, anxiety/distress, sleep difficulties, fatigue, and lack of appetite) using a 0-10 numeric rating scale, with 10 indicating a higher severity, in daily diary format.
change in mean peak severity for sleep difficulties across all three cycles | up to 11 weeks
  Subjects will complete a self-report Symptom Inventory Diary during each Study Cycle starting at Day 0 and continuing to Day 6. Subjects will rate the severity of seven symptoms (nausea, vomiting, pain, anxiety/distress, sleep difficulties, fatigue, and lack of appetite) using a 0-10 numeric rating scale, with 10 indicating a higher severity, in daily diary format.
change in mean peak severity for lack of appetite across all three cycles | up to 11 weeks
  Subjects will complete a self-report Symptom Inventory Diary during each Study Cycle starting at Day 0 and continuing to Day 6. Subjects will rate the severity of seven symptoms (nausea, vomiting, pain, anxiety/distress, sleep difficulties, fatigue, and lack of appetite) using a 0-10 numeric rating scale, with 10 indicating a higher severity, in daily diary format.
the number of participants who found the aromatherapy acceptable | up to 11 weeks
  The following questions will be asked of the subjects to obtain qualitative feedback to further evaluate acceptability of the aromatherapy inhalers: 1) What two things did you like about your aromatherapy inhaler?; 2) What two things did subjects dislike about the aromatherapy inhaler?; 3) Was the aromatherapy inhaler easy to use?; 4) Did subjects feel that the aromatherapy inhaler reduced symptoms from chemotherapy? Please circle the symptoms that seemed to be helped the most.; 5) Would the subject use this aromatherapy inhaler again in the future?; 6) Would the subject recommend this aromatherapy inhaler to others?; 7) What word or statement would the subject use to describe their experience during this clinical trial?; and 8) What intervention arm do subjects think they were in? All of these data will help determine if the aromatherapy inhalers and scents are acceptable and feasible to use for in cancer subjects during chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Ryan, PhD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester Medical Center, Wilmot Canter Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lua PL, Zakaria NS. A brief review of current scientific evidence involving aromatherapy use for nausea and vomiting. J Altern Complement Med. 2012 Jun;18(6):534-40. doi: 10.1089/acm.2010.0862. PMID 22784340
- [Background] Stringer J, Donald G. Aromasticks in cancer care: an innovation not to be sniffed at. Complement Ther Clin Pract. 2011 May;17(2):116-21. doi: 10.1016/j.ctcp.2010.06.002. PMID 21457903
- [Background] Bradley BF, Starkey NJ, Brown SL, Lea RW. Anxiolytic effects of Lavandula angustifolia odour on the Mongolian gerbil elevated plus maze. J Ethnopharmacol. 2007 May 22;111(3):517-25. doi: 10.1016/j.jep.2006.12.021. Epub 2006 Dec 27. PMID 17289317
- [Background] de Almeida RN, Motta SC, de Brito Faturi C, Catallani B, Leite JR. Anxiolytic-like effects of rose oil inhalation on the elevated plus-maze test in rats. Pharmacol Biochem Behav. 2004 Feb;77(2):361-4. doi: 10.1016/j.pbb.2003.11.004. PMID 14751465
- [Background] Dyer J, Cleary L, Ragsdale-Lowe M, McNeill S, Osland C. The use of aromasticks at a cancer centre: a retrospective audit. Complement Ther Clin Pract. 2014 Nov;20(4):203-6. doi: 10.1016/j.ctcp.2013.11.006. Epub 2013 Nov 28. PMID 25486854
- [Background] Boehm K, Bussing A, Ostermann T. Aromatherapy as an adjuvant treatment in cancer care--a descriptive systematic review. Afr J Tradit Complement Altern Med. 2012 Jul 1;9(4):503-18. doi: 10.4314/ajtcam.v9i4.7. eCollection 2012. PMID 23983386
- [Background] Lillehei AS, Halcon LL. A systematic review of the effect of inhaled essential oils on sleep. J Altern Complement Med. 2014 Jun;20(6):441-51. doi: 10.1089/acm.2013.0311. Epub 2014 Apr 10. PMID 24720812
- [Background] Wood LJ, Nail LM, Gilster A, Winters KA, Elsea CR. Cancer chemotherapy-related symptoms: evidence to suggest a role for proinflammatory cytokines. Oncol Nurs Forum. 2006 May 3;33(3):535-42. doi: 10.1188/06.ONF.535-542. PMID 16676010
- [Background] Jordan K, Gralla R, Jahn F, Molassiotis A. International antiemetic guidelines on chemotherapy induced nausea and vomiting (CINV): content and implementation in daily routine practice. Eur J Pharmacol. 2014 Jan 5;722:197-202. doi: 10.1016/j.ejphar.2013.09.073. Epub 2013 Oct 21. PMID 24157984
- [Background] Marx WM, Teleni L, McCarthy AL, Vitetta L, McKavanagh D, Thomson D, Isenring E. Ginger (Zingiber officinale) and chemotherapy-induced nausea and vomiting: a systematic literature review. Nutr Rev. 2013 Apr;71(4):245-54. doi: 10.1111/nure.12016. Epub 2013 Mar 13. PMID 23550785
- [Background] Ryan JL. Treatment of Chemotherapy-Induced Nausea in Cancer Patients. Eur Oncol. 2010;6(2):14-16. doi: 10.17925/eoh.2010.06.02.14. PMID 21984886
- [Background] Ryan JL, Heckler CE, Roscoe JA, Dakhil SR, Kirshner J, Flynn PJ, Hickok JT, Morrow GR. Ginger (Zingiber officinale) reduces acute chemotherapy-induced nausea: a URCC CCOP study of 576 patients. Support Care Cancer. 2012 Jul;20(7):1479-89. doi: 10.1007/s00520-011-1236-3. Epub 2011 Aug 5. PMID 21818642
- [Background] Hines S, Steels E, Chang A, Gibbons K. Aromatherapy for treatment of postoperative nausea and vomiting. Cochrane Database Syst Rev. 2012 Apr 18;(4):CD007598. doi: 10.1002/14651858.CD007598.pub2. PMID 22513952
- [Background] Lien HC, Sun WM, Chen YH, Kim H, Hasler W, Owyang C. Effects of ginger on motion sickness and gastric slow-wave dysrhythmias induced by circular vection. Am J Physiol Gastrointest Liver Physiol. 2003 Mar;284(3):G481-9. doi: 10.1152/ajpgi.00164.2002. PMID 12576305
- [Background] Bone ME, Wilkinson DJ, Young JR, McNeil J, Charlton S. Ginger root--a new antiemetic. The effect of ginger root on postoperative nausea and vomiting after major gynaecological surgery. Anaesthesia. 1990 Aug;45(8):669-71. doi: 10.1111/j.1365-2044.1990.tb14395.x. PMID 2205121
- [Background] Grontved A, Brask T, Kambskard J, Hentzer E. Ginger root against seasickness. A controlled trial on the open sea. Acta Otolaryngol. 1988 Jan-Feb;105(1-2):45-9. doi: 10.3109/00016488809119444. PMID 3277342
- [Background] Kim S, Kim HJ, Yeo JS, Hong SJ, Lee JM, Jeon Y. The effect of lavender oil on stress, bispectral index values, and needle insertion pain in volunteers. J Altern Complement Med. 2011 Sep;17(9):823-6. doi: 10.1089/acm.2010.0644. Epub 2011 Aug 19. PMID 21854199
- [Background] Goes TC, Antunes FD, Alves PB, Teixeira-Silva F. Effect of sweet orange aroma on experimental anxiety in humans. J Altern Complement Med. 2012 Aug;18(8):798-804. doi: 10.1089/acm.2011.0551. Epub 2012 Jul 31. PMID 22849536
- [Background] Jafarzadeh M, Arman S, Pour FF. Effect of aromatherapy with orange essential oil on salivary cortisol and pulse rate in children during dental treatment: A randomized controlled clinical trial. Adv Biomed Res. 2013 Mar 6;2:10. doi: 10.4103/2277-9175.107968. Print 2013. PMID 23930255
- [Background] Ndao DH, Ladas EJ, Cheng B, Sands SA, Snyder KT, Garvin JH Jr, Kelly KM. Inhalation aromatherapy in children and adolescents undergoing stem cell infusion: results of a placebo-controlled double-blind trial. Psychooncology. 2012 Mar;21(3):247-54. doi: 10.1002/pon.1898. Epub 2010 Dec 27. PMID 22383266
- [Background] Habashy RR, Abdel-Naim AB, Khalifa AE, Al-Azizi MM. Anti-inflammatory effects of jojoba liquid wax in experimental models. Pharmacol Res. 2005 Feb;51(2):95-105. doi: 10.1016/j.phrs.2004.04.011. PMID 15629254
- [Background] Kohara H, Miyauchi T, Suehiro Y, Ueoka H, Takeyama H, Morita T. Combined modality treatment of aromatherapy, footsoak, and reflexology relieves fatigue in patients with cancer. J Palliat Med. 2004 Dec;7(6):791-6. doi: 10.1089/jpm.2004.7.791. PMID 15684846
- [Background] Pazyar N, Yaghoobi R, Ghassemi MR, Kazerouni A, Rafeie E, Jamshydian N. Jojoba in dermatology: a succinct review. G Ital Dermatol Venereol. 2013 Dec;148(6):687-91. PMID 24442052
- [Background] Axel R. The molecular logic of smell. Sci Am. 1995 Oct;273(4):154-9. doi: 10.1038/scientificamerican1095-154. PMID 7481719
- [Background] Borm GF, Fransen J, Lemmens WA. A simple sample size formula for analysis of covariance in randomized clinical trials. J Clin Epidemiol. 2007 Dec;60(12):1234-8. doi: 10.1016/j.jclinepi.2007.02.006. Epub 2007 Jun 6. PMID 17998077
- [Background] Little R, Yau L. Intent-to-treat analysis for longitudinal studies with drop-outs. Biometrics. 1996 Dec;52(4):1324-33. PMID 8962456
- See also: Aromatherapy NAoH. Explore Aromatherapy: Safety Raleigh, NC2015 — http://naha.org/explore-aromatherapy/safety/